CLINICAL TRIAL: NCT07006376
Title: Investigation of Thoracolumbar Fascia Thickness, Trunk Flexibility and Manual Dexterity in Parkinson's Disease Patients
Brief Title: Thoracolumbar Fascia Thickness in Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Büşra Seçkinoğulları Korkusuz, Principal Investigator, Ankara University
Other Study IDs: E-59394181-604.01-112208
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to examine thoracolumbar fascia thickness, trunk flexibility, trunk control and upper extremity skills in Parkinson's disease patients. Patients between the ages of 55-80 who have been diagnosed with Parkinson's disease by a neurologist and healthy individuals with similar demographic characteristics will be included in the study as a control group. Demographic information of the individuals will be recorded and clinical evaluations will be made. Staging of Parkinson's patients will be done with the Modified Hoehn and Yahr Scale (MHRS), and disease severity will be done with the Unified Parkinson's Disease Rating Scale (UPDRS). Thoracolumbar fascia thickness of individuals in both groups will be evaluated with ultrasonography, trunk flexibility with the Active Trunk Range of Motion Assessment and Sit-Reach test, trunk functions with the Trunk Impairment Scale, and manual skills with the Purdue Pegboard Test.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 80
* Mini Mental State Examination (MMSE) score between 24 and 30
* Diagnosed with Parkinson's by a neurologist
* MH&Y stage 2-3

Exclusion Criteria:

* Inability to communicate verbally
* Use of walking aids
* Elderly people with severe visual impairment, neurological disorders and/or congestive heart failure
* Older adults in whom exercise is not recommended.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Ultrasonography Measurement | Baseline
  The thickness of the Thoracolumbar Fascia will be measured by ultrasonography at the level of the L3 lumbar vertebra and using a predefined standard protocol.
Range of Motion Assessment | Baseline
  Active trunk ranges of motion will be assessed during flexion/extension, rotation, and lateral flexion using a universal goniometer.
Sit and Reach Test | Baseline
  For this test, a tape measure will be fixed to a table at the exact level of the subjects' feet. Subjects will sit in front of the table with bare feet and legs straight. Then, they will slowly extend forward as far as possible, keeping their hands together and without bending their knees. During this extension, attention will be paid to the subjects' straight backs and to avoid sudden movements.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla Fil Balkan, Assoc Prof, Study Chair — Hacettepe University; Gül Yalçın Çakmaklı, Assoc Prof, Study Chair — Hacettepe University; Süleyman Korkusuz, Assist.Prof, Study Chair — Atılım University; Büşra Seçkinoğulları Korkusuz, PhD, Principal Investigator — Ankara University
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] De Coninck K, Hambly K, Dickinson JW, Passfield L. Measuring the morphological characteristics of thoracolumbar fascia in ultrasound images: an inter-rater reliability study. BMC Musculoskelet Disord. 2018 Jun 1;19(1):180. doi: 10.1186/s12891-018-2088-5. PMID 29859080
- [Background] Yerli S, Yinanc SB, Yagci G, Erbahceci F, Ozcakar L. Thoracolumbar fascia and chronic low back pain in idiopathic lumbar scoliosis: an ultrasonographic study. Eur Spine J. 2024 Jun;33(6):2469-2475. doi: 10.1007/s00586-024-08266-x. Epub 2024 Apr 23. PMID 38653872